CLINICAL TRIAL: NCT00759356
Title: A Single-Dose, 2-Period, 2-Treatment, 2-Way Crossover Study Comparing the Bioavailability of a Morphine Sulfate Sustained Release Capsule 1 x 200mg to KADIAN 2 x 100mg Capsules Under Fed Conditions
Brief Title: Comparison of One Morphine Sulfate Sustained-Release 200mg Capsule With Two 100 mg KADIAN Capsules Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Daniel V. Freeland, DO, CEDRA Clinical Research, LLC
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20-700-1N
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2009-09-01 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: bioavailability; KADIAN; 200 mg; morphine sulfate sustained release capsules; 100 mg; fed conditions
MeSH Terms: interventions — Morphine

ARMS (2):
- 1 (Other): Treatment A (test product) followed by Treatment B (reference product)
  Interventions: Drug: morphine sulfate sustained-release capsules; Drug: KADIAN
- 2 (Other): Treatment B (reference product) followed by Treatment A (test product)
  Interventions: Drug: morphine sulfate sustained-release capsules; Drug: KADIAN

INTERVENTIONS:
Drug: morphine sulfate sustained-release capsules — 1 x 200 mg, single-dose capsule
  Other Names: Treatment A; Test Product
Drug: KADIAN — 2 x 100 mg, single-dose capsule
  Other Names: Treatment B; Reference Product

SUMMARY:
The objective of this single-dose, open-label, randomized, two-period crossover study was to compare the rate of absorption and oral bioavailability of a test formulation of morphine sulfate 200 mg sustained-release capsules manufactured by Alpharma Branded Products Division Inc. to an equivalent oral dose of the commercially available reference product, KADIAN 2 x 100 mg capsules manufactured by Alpharma Branded Products Division Inc. when administered under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a male or non-pregnant, non-breast-feeding female.
* Subject must be between 18 and 50 years of age inclusive.
* Subject's body weight should be within +/- 15% of the ideal body weight for their height and estimated frame based on the Metropolitan Life Insurance Company Table and weigh a minimum of 50 kg (110 lbs).
* Female subjects - not surgically sterile or at least two years postmenopausal - must agree to utilize one of the following forms of contraception, if sexually active with a male partner, from screening through completion of the study. Approved forms of contraception are abstinence, hormonal (oral, implant, transdermal or injection), double barrier (condom and diaphragm with spermicide), IUD, or vasectomized partner (6 months minimum).
* Subject must voluntarily consent to participate in this study and provide their written informed consent prior to completion of any study-specific procedures.
* Subject is willing and able to remain in the study unit for the entire duration of each confinement period and return to the study site for any outpatient visits.

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic or psychiatric disease or any other condition which, in the opinion of the Investigator would jeopardize the safety of the subject or the validity of the study results.
* Has a clinically significant abnormal finding on the physical exam, medical history or clinical laboratory results at screening.
* History or presence of allergic or adverse response to the study drug or related drugs.
* Has been on a significantly abnormal diet during the four weeks preceding the first dose of study medication.
* Has donated blood or plasma within 30 days prior to the first dose of study medication.
* Has participated in another clinical trial within 30 days prior to first dose of study medication.
* Has used any over-the-counter (OTC) medication including vitamins, within 7 days prior to the first dose of study medication without evaluation and approval by the study investigator.
* Has used any prescription medication, except hormonal contraceptive or hormonal replacement therapy, within 7 days prior to the first dose of study medication without evaluation and approval by the study investigator.
* Has been treated with any known enzyme altering drugs such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of study medication.
* Has smoked or used tobacco products within 60 days prior to the first dose of study medication.
* Has a history of substance abuse (including alcohol) in the past 5 years.
* Is a female with a positive pregnancy test result.
* Has a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates).
* Has had a positive test for, or has been treated for hepatitis B, hepatitis C or HIV.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2004-08; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel V. Freeland, DO, Principal Investigator — CEDRA Clinical Research, LLC
Locations (1):
- CEDRA Clinical Research, LLC, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Wash out period of at least 7 days.
Groups:
- Period 1: Treatment A or B: Treatment A (test product) followed by Treatment B (reference product)
- Period 2: Treatment A or B: Treatment B (reference product) followed by Treatment A (test product)
Period: Overall Study
Arm/Group | Period 1: Treatment A or B | Period 2: Treatment A or B
Started | 18 | 18
Completed | 17 | 15
Not Completed | 1 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Subject was unable to return | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Period 1: Treatment A or B | Period 2: Treatment A or B | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.5 (7.5) | 33.9 (6.3) | 31.7 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Mean Maximum Plasma Morphine Concentration
Time Frame: 0 (predose), and 2,4,6,6.5,7,7.5,8,8.5,9,9.5,10,12,18,24,30,36,48 hrs post dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Morphine Sulfate SR 200 mg Capsule | KADIAN® 200 mg Capsule
Number analyzed (Participants) | 28 | 28
ng/mL | 37.3 (15.8) | 32.8 (11.6)
Statistical Analysis 1: Comparison: Morphine Sulfate SR 200 mg Capsule vs KADIAN® 200 mg Capsule; Test type: Non-Inferiority or Equivalence — The 90% confidence intervals for the ratios (test/reference) of the least squares means of the non-transformed parameters Cmax, AUClast, AUCinf, Tmax, λz, and T1/2, were calculated; ANOVA; Mean ratio = 109.8, 90% CI [95.3 to 126.5]

2. Secondary Outcome: Time of Maximum Plasma Morphine Concentration
Time Frame: 0 (predose), and 2,4,6,6.5,7,7.5,8,8.5,9,9.5,10,12,18,24,30,36,48 hrs post dose
Measure: Median (Full Range); unit: hr
Arm/Group | Morphine Sulfate SR 200 mg Capsule | KADIAN® 200 mg Capsule
Number analyzed (Participants) | 28 | 28
hr | 12.00 (4.95) [8.00 to 24.00] | 12.00 (6.25) [8.00 to 30.00]

3. Secondary Outcome: Area Under the Curve to the Last Measurable Time Point for Plasma Morphine
Time Frame: 0 (predose), and 2,4,6,6.5,7,7.5,8,8.5,9,9.5,10,12,18,24,30,36,48 hrs post dose
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Morphine Sulfate SR 200 mg Capsule | KADIAN® 200 mg Capsule
Number analyzed (Participants) | 28 | 28
hr*ng/mL | 691.3 (196.0) | 674.1 (169.7)
Statistical Analysis 1: Comparison: Morphine Sulfate SR 200 mg Capsule vs KADIAN® 200 mg Capsule; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; mean ratio = 101.5, 90% CI [95.6 to 107.9]

4. Secondary Outcome: Area Under the Curve to Infinity for Plasma Morphine
Time Frame: 0 (predose), and 2,4,6,6.5,7,7.5,8,8.5,9,9.5,10,12,18,24,30,36,48 hrs post dose
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Morphine Sulfate SR 200 mg Capsule | KADIAN® 200 mg Capsule
Number analyzed (Participants) | 28 | 28
hr*ng/mL | 800.3 (220.9) | 789.2 (237.5)
Statistical Analysis 1: Comparison: Morphine Sulfate SR 200 mg Capsule vs KADIAN® 200 mg Capsule; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; log-transformation; mean ratio = 101.7, 90% CI [95.9 to 107.9]

ADVERSE EVENTS:
Arm/Group | Arm 1: Treatment A Followed by Treatment B | Arm 2: Treatment B Followed by Treatment A
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 11 | 9
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Arm 1: Treatment A Followed by Treatment B | Arm 2: Treatment B Followed by Treatment A
Somnolence (Nervous system disorders) | 3/18 (3) | 1/18 (1)
Abdominal Pain (Gastrointestinal disorders) | 4/18 (4) | 1/18 (2)
Nausea (Gastrointestinal disorders) | 7/18 (10) | 8/18 (9)
Headache (Nervous system disorders) | 2/18 (5) | 6/18 (6)
Vomiting (Gastrointestinal disorders) | 3/18 (3) | 3/18 (3)
Fatigue (General disorders) | 1/18 (1) | 0/18 (0)
Flushing (Vascular disorders) | 1/18 (1) | 0/18 (0)
Rhinitis (Infections and infestations) | 1/18 (1) | 0/18 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1/18 (1) | 0/18 (0)
Tremors (Nervous system disorders) | 1/18 (1) | 0/18 (0)
Abdominal Distention (Gastrointestinal disorders) | 1/18 (1) | 0/18 (0)
Anxiety (Psychiatric disorders) | 0/18 (0) | 1/18 (1)
Dyspepsia (Gastrointestinal disorders) | 0/18 (0) | 1/18 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0/18 (0) | 1/18 (1)
Diarrhea (Gastrointestinal disorders) | 0/18 (0) | 2/18 (2)
Chills (General disorders) | 0/18 (0) | 1/18 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No